CLINICAL TRIAL: NCT07387666
Title: A Prospective, Open-label Phase 0 Single-center Study to Assess the Effect of Acetadote on Metabolism in Newly Diagnosed Glioblastoma
Brief Title: Imaging Acetadote Metabolism in Glioblastoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Evan Noch, ASSISTANT PROFESSOR, Neurology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU20250529; SCCC-07325
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma; GBM
MeSH Terms: conditions — Glioblastoma | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acetadote 150 mg/kg IV (Experimental): Acetadote will be administered twice during this study: first before undergoing magnetic resonance spectroscopy (MRS) on Day 1 and second before undergoing surgical resection, which will take place between Days 2-21. Acetadote will be administered at a dose of 150 mg/kg IV over 60 minutes.
  Interventions: Drug: Acetadote

INTERVENTIONS:
Drug: Acetadote — Acetadote 150 mg/kg in 500 cc 5% dextrose IV over 1 hour

SUMMARY:
This goal of this clinical trial is to evaluate how Acetadote affects metabolism in patients with glioblastoma. Drugs like Acetadote, which affect the level of damage in a cell (oxidative stress), may impact brain tumor metabolism and slow the growth of brain tumors.

The investigators are evaluating how Acetadote affects glioblastoma metabolism by using MRI-based methods and by determining the changes in metabolism in brain tumor tissue resected from patients with a new diagnosis of glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Glioblastoma
* 2. Newly diagnosed with no prior surgery, radiation, chemotherapy, or other tumor-treating agent
* 3. Age ≥18 years
* 4. KPS > 70
* 5. Adequate organ and marrow function as defined below:
* - Bilirubin ≤1.5 times upper limit of normal
* - AST and ALT ≤ 3 times ULN
* - Creatinine ≤ 1.5 x ULN and/or GFR ≤ 60 mL/min
* -ANC ≥ 1000 cells/ul
* - Platelet ≥ 100,000/ul
* - Hemoglobin ≥ 9 g/dl
* 6. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 7 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* 6a. A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* - Has not undergone a hysterectomy or bilateral oophorectomy; or
* - Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* 7. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* 1.Chemotherapy, radiotherapy, or other cancer therapy within 4 weeks prior to starting study treatment.
* 2. Subjects must have recovered from prior treatment-related toxicities to grade 2 or baseline (excluding alopecia and clinically stable toxicities requiring ongoing medical management, such as hypothyroidism from prior immune checkpoint inhibitor treatment).
* 3. Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
* 4. Brain metastases
* 5. History of allergic or hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to Acetadote.
* 6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* 7. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of Acetadote on glioblastoma metabolism as measured by MRS. | Day 1 and up to 21 days from Day 1
  The effect of Acetadote on glioblastoma metabolism will be assessed by measuring cysteine, glutathione, and lactate in glioblastoma through MRS.

SECONDARY OUTCOMES:
To determine the effect of Acetadote on glioblastoma metabolism in resected tumor tissue as measured by LCMS | Day 1 and up to 21 days from Day 1
  The effect of Acetadote on glioblastoma metabolism in resected tumor tissue will be measured by Liquid chromatography-mass spectrometry (LCMS).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No